CLINICAL TRIAL: NCT05886634
Title: A Phase II Study of Adenosine Receptor (A2A and A2B) Inhibition (AB928) in Combination With Anti-PD-1 Therapy (AB122) in Patients With Advanced Dedifferentiated Liposarcoma
Brief Title: A Study of Etrumadenant and Zimberelimab in People With Dedifferentiated Liposarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-277
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Dedifferentiated Liposarcoma; Soft Tissue Sarcoma; Sarcoma,Soft Tissue; Sarcoma; Recurrent Dedifferentiated Liposarcoma; Unresectable Dedifferentiated Liposarcoma; Metastatic Dedifferentiated Liposarcoma
Keywords: Dedifferentiated Liposarcoma; Recurrent Dedifferentiated Liposarcoma; Unresectable Dedifferentiated Liposarcoma; Metastatic Dedifferentiated Liposarcoma; Soft Tissue Sarcoma; Sarcoma, Soft Tissue; Sarcoma; DDLPS; Memorial Sloan Kettering Cancer Center; 22-277
MeSH Terms: conditions — Liposarcoma; Sarcoma | interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants With Dedifferentiated Liposarcoma/DDLPS (Experimental): Participants will have a diagnosis of recurrent or metastatic Dedifferentiated Liposarcoma/DDLPS
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab

INTERVENTIONS:
Drug: Etrumadenant — Will be administered PO daily for 24 weeks
Drug: Zimberelimab — Will be administered IV every 2 weeks for 24 weeks

SUMMARY:
Participants will have a diagnosis of dedifferentiated liposarcoma (DDLS) that has spread beyond its original location (advanced). In addition, their DDLS either has come back after treatment (recurrent), has spread to different parts of your body (metastatic), or is unable to be removed surgically (unresectable). The purpose of this study is to find out whether the combination of etrumadenant and zimberelimab is an effective treatment for people with advanced DDLS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent, unresectable, or metastatic DDLPS

  * The definition of recurrent disease is a patient with a primary tumor that has been successfully resected, but has recurred after primary surgery
  * Any number of prior systemic therapies will be allowed
* Age ≥ 18 years at the time of informed consent
* Willing and able to provide written informed consent/assent for the trial
* Willing to comply with treatment protocol
* Adequate performance status: Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1/Karnofsky Performance Status (KPS) 70-100%
* Presence of measurable disease per RECIST v1.1

  o Target lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression
* QTc ≤ 480 msec using Fredericia's QT correction formula
* Adequate organ function determined within 2 weeks of treatment initiation, defined as follows:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1,500/mm3 (1.0 x 109/L)
  * Platelet count ≥ 75,000/mm3 (50 x 109/L)
  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) OR direct bilirubin ≤ ULN for a patient with total bilirubin level > 1.5 x ULN
  * Aspartate aminotransferase (AST) ≤ 2.5 x ULN OR ≤ 5 x ULN for patients with liver metastases
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN OR ≤ 5 x ULN for patients with liver metastases
  * Alkaline phosphatase < 5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or a measured or calculated creatinine clearancea

    ≥ 60 mL/min for a patient with creatinine levels > 1.5 x institutional ULN (Note: Creatinine clearance need not be determined if the baseline serum creatinine is within normal limits. GFR can also be used in place of creatinine or CrCl)
  * International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT and PTT is within therapeutic range of intended use of anticoagulants
* For female patients of childbearing potential, negative serum pregnancy test at screening visit and within 72 h prior to the first dose of study medication

aCreatinine clearance should be calculated per institutional standard.

Contraception Requirements

Female participants of reproductive potential and male participants with female partners of reproductive potential are required to use highly effective contraceptive measures from the first dose of study treatment until 30 days after the last dose of etrumadenant or 90 days after the last dose of zimberelimab, whichever is longer.

* A female participant (or female partner of a male participant) is considered fertile following menarche and until becoming post-menopausal unless permanently sterile.

  * Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
  * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
* A man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy

Highly effective contraception is defined as use of one or more methods that result in a low failure rate (i.e., less than 1%). Highly effective contraceptive measures include:

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
* Progestogen only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
* Intrauterine device
* Intrauterine hormone-releasing system in combination with a barrier method (preferably male condom)
* Surgical sterilization

  * Female participant or female partner of the male participant has undergone bilateral tubal ligation
  * Male participant is vasectomized (with documented medical confirmation of surgical success) and is the sole sexual partner of a female with reproductive potential
* Complete sexual abstinence defined as refraining from heterosexual intercourse during the entire period of risk associated with study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant

To ensure proper birth control, female participants who use hormonal contraception should use an efficient barrier contraceptive (condom plus spermicide). Additionally, male participants, when having sexual intercourse with a female of reproductive potential, should use an efficient barrier contraceptive (condom plus spermicide); the respective partner should also use an additional efficient contraceptive method (e.g., oral pills, intrauterine device, or diaphragm, and spermicide).

Exclusion Criteria:

Patients who fulfil any of the following criteria are not eligible for admission to the study:

* Prior treatment with systemic PD-1 or PD-L1 inhibitor
* Prior treatment with an agent targeting the adenosine pathway
* Have a concurrent unrelated malignancy that requires active treatment

  o Patients with concurrent malignancies of a different tumor whose natural history or treatment will likely not interfere with the safety or efficacy assessment of the investigational drug will be eligible
* Uncontrolled intercurrent illness including active infection requiring systemic therapy or symptomatic congestive heart failure within the past 6 months
* Has known active central nervous system (CNS) metastases

  * Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to study Day 1 and return to baseline of neurologic symptoms), and have no evidence of new or enlarging brain metastases. This exception does not include sarcomatous meningitis, which is excluded regardless of clinical stability.
  * Patients must be on a stable or decreasing corticosteroid dose at the time of study entry; patients who require escalating doses of corticosteroids for the treatment of CNS metastases will be excluded.
* Shows evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 14 days prior to enrollment. However, in the setting of non-immune mediated indications for use, chronic/active low dose steroid use may be permitted at the discretion of the principal investigator.
* Has a known infection with HIV AND

  * CD4+ T-cell (CD4+) counts < 350 cells/uL
  * An opportunistic infection within the prior 12 months
* Has a known active infection with hepatitis B or hepatitis C

  * Chronic carriers of HBV infection (HBsAg-positive, undetectable or low HBV DNA, and normal ALT) or individuals who have serologic evidence of a resolved prior HBV infection (i.e., HBsAg-negative and anti-HBc-positive) may be eligible if suppressive antiviral therapy can be safely administered.
  * Patients who have completed curative antiviral treatment for HCV and have a viral load below the limit of quantification will be eligible (e.g. a patient who is HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution)
* Has a known history of active tuberculosis infection
* Has history or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in the past 2 years.

Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease.

* For female subjects, is pregnant or breast-feeding, or planning to become pregnant
* For male subjects, is planning to father a child within the projected duration of the trial, starting with the pre-screening or screening visit, during study treatment and through 4 months after the last cycle of treatment
* For patients of childbearing potential, is unwilling to use acceptable method(s) of effective contraception during study treatment and through 4 months after the last cycle of treatment. (Women not of childbearing potential are defined as: post-menopausal [age > 55 years with cessation of menses for 12 or more months or less than 55 years but not spontaneous menses for at least 2 years or less than 55 years and spontaneous menses within the past 1 year, but currently amenorrhoeic (e.g., spontaneous or secondary to hysterectomy), and with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved] or who have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.)
* Underwent prior chemotherapy, radiotherapy, biological cancer therapy, targeted small molecule therapy, or major surgery within 4 weeks (or 5 half-lives, whichever is shorter) prior to study Day 1 or has not recovered (i.e., to CTCAE ≤ grade 1 or at baseline) from adverse events due to previously administered therapy. Patients with ≤ grade 2 neuropathy and alopecia are an exception and may qualify for the study. If patients received major surgery, they must have recovered adequately prior to starting therapy.
* Is currently participating and receiving study therapy with another investigational device or study drug or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks (or 5 half-lives, whichever is shorter) of the first dose of treatment
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Prior organ transplantation, including allogeneic stem-cell transplant
* Due to the potential risk for drug-drug interactions with etrumadenant, participants must not have had:

  * Treatment with known BCRP substrates with a narrow therapeutic window, administered orally (e.g., prazosin, rosuvastatin) within 4 weeks or 5 half-lives of the drug (whichever is shorter) prior to initiation of and throughout study treatment
  * Treatment with known P-gp substrates with a narrow therapeutic window, administered orally (e.g., digoxin) within 4 weeks or 5 half-lives of the drug (whichever is shorter) prior to initiation of study treatment
  * Treatment with known strong CYP3A4 inducers (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) and strong CYP3A4 inhibitors (e.g., clarithromycin, grapefruit juice, itraconazole, ketoconazole, posaconazole, telithromycin, and voriconazole) within 4 weeks or 5 half lives of the drug (whichever is shorter) prior to initiation of study treatment
  * Refer to the following for more examples of relevant substrates, inhibitors, and inducers with the potential for drug-drug interactions with etrumadenant: https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers
* Any gastrointestinal condition that would preclude the use of oral medications (e.g., difficulty swallowing, nausea, vomiting, or malabsorption)
* History of severe allergic reactions to chimeric or humanized antibodies or fusion protein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2027-05-23 (Estimated); Study Completion 2027-05-23 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 24 weeks
  To estimate the overall response rate (CR + PR per RECIST 1.1) to etrumadenant combined with zimberelimab at 24 weeks in patients with advanced Dedifferentiated Liposarcoma/DDLPS

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York